CLINICAL TRIAL: NCT07303205
Title: Predictive Value of the Preoperative ROX Index for Early Postoperative Hypoxemia in Bariatric Surgery Patients: A Prospective Observational Cohort Study
Brief Title: Preoperative ROX Index and Postoperative Hypoxemia in Bariatric Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Istinye University
Other Study IDs: erkan rox indeksi
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Preoperative ROX Index Assessment — Participants will undergo a preoperative assessment including measurement of the ROX index (SpO₂/FiO₂ divided by respiratory rate) before bariatric surgery. No treatment or study-related intervention will be applied; all perioperative care will follow routine clinical practice.

SUMMARY:
This prospective observational study evaluates whether the preoperative ROX index can predict early postoperative hypoxemia in patients undergoing bariatric surgery. Preoperative ROX measurements, along with ARISCAT and STOP-Bang scores, will be assessed for their association with hypoxemia occurring within the first 12 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Scheduled for elective bariatric surgery (laparoscopic sleeve gastrectomy or Roux-en-Y gastric bypass)
* Body mass index (BMI) ≥ 35 kg/m²
* ASA physical status I-III
* Able and willing to provide written informed consent

Exclusion Criteria:

* Acute respiratory failure, pneumonia, or active pulmonary infection
* Receiving oxygen therapy or respiratory support (nasal cannula, CPAP, BiPAP, or high-flow oxygen) preoperatively
* Preoperative SpO₂ < 88% on room air
* Significant cardiac arrhythmia, severe heart failure (NYHA class III-IV), or hemodynamic instability
* Pregnancy, active malignancy, or current immunosuppressive therapy
* Inability to complete postoperative follow-up or early discharge before 12-hour assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients scheduled for elective bariatric surgery, including laparoscopic sleeve gastrectomy and Roux-en-Y gastric bypass. All participants are obese (BMI ≥ 35 kg/m²) and evaluated preoperatively in the anesthesia clinic prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Early Postoperative Hypoxemia | Postoperative 0-12 hours
  Hypoxemia defined as SpO₂ < 92% or new oxygen requirement within the first postoperative hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

REFERENCES:
- [Result] Helmy MA, Mostafa MS, Saber AT, Ali MA, Milad LM. Erector Spinae Plane Block and its Impact on Postoperative Diaphragmatic Dysfunction in Morbidly Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy: A Double-Blind Randomized Control Trial. Obes Surg. 2025 Dec;35(12):5228-5236. doi: 10.1007/s11695-025-08337-y. Epub 2025 Nov 4. PMID 41188672
- [Result] Wang X, Guo K, Sun J, Yang Y, Wu Y, Tang X, Xu Y, Chen Q, Zeng S, Wang L, Liu S. Semirecumbent Positioning During Anesthesia Recovery and Postoperative Hypoxemia: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2416797. doi: 10.1001/jamanetworkopen.2024.16797. PMID 38941098
- [Result] Lee S, Hong H, Cho H, Lee SW, You AH, Kang HY, Park SW, Kim MK, Choi JH. Association between preoperative oxygen reserve index and postoperative pulmonary complications: a prospective observational study. Korean J Anesthesiol. 2025 Jun;78(3):224-235. doi: 10.4097/kja.24420. Epub 2025 Feb 17. PMID 40468628